CLINICAL TRIAL: NCT00664755
Title: Menstrual Cycle Effects on Smoking Cessation and Cue Reactivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Kevin Gray, MD, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P50DA016511 (NIH)
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Results first posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-04

CONDITIONS: Nicotine Dependence
Keywords: Menstrual Cycle effects; Cue Reactivity; Smoking Cessation; Impulsivity
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Impulsive Behavior | interventions — Varenicline; Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Experimental): Participant randomized to receive active varenicline and placebo transdermal nicotine patch.
  Interventions: Drug: varenicline
- Transdermal Nicotine Patch (Active Comparator): Participant randomized to receive active transdermal nicotine patch and placebo varenicline.
  Interventions: Device: transdermal nicotine patch

INTERVENTIONS:
Drug: varenicline — Day -7 thru -5: 0.5mg QD Day -4 thru -1: 0.5mg BID Day 0 onward: 1.0mg BID
  Varenicline is taken for a duration of 4 weeks in this study.
  Other Names: Chantix
  Arms: Varenicline
Device: transdermal nicotine patch — Weeks 0-3: 21mg patch
  Transdermal nicotine patch is used for a duration of 3 weeks in this study.
  Other Names: Nicoderm CQ
  Arms: Transdermal Nicotine Patch

SUMMARY:
This is a brief smoking cessation trial in women, comparing transdermal nicotine patch (TNP) versus varenicline.

DETAILED DESCRIPTION:
This component builds directly upon the results of the previously funded project in systematically investigating the impact of short-term ovarian hormone fluctuation on females as they try to quit smoking with the aid of either transdermal nicotine patch (TNP) or varenicline. Each participant will receive a standardized impulsivity evaluation and a laboratory-based cue reactivity assessment before the initiation of smoking cessation. Progesterone and estrogen levels will be measured at each of nine visits, thereby providing an index of reproductive hormone variation over the course of each participant's quit attempt. This novel approach of integrating a human laboratory cue reactivity paradigm directly with a treatment outcome study will permit us to assess whether or not smoking cue reactivity has predictive utility with respect to cessation outcome. Subjects will be randomized to receive one of two active pharmacotherapeutic interventions for smoking cessation: TNP vs. varenicline in a randomized, single-blind, double dummy design. While TNP has demonstrated modest efficacy in improving smoking cessation outcomes, there is some evidence that its efficacy may be more robust in men as compared to women. This project will provide important information about a) the impact of ovarian hormone levels on smoking cessation outcomes, b) the relationship between smoking cue reactivity and smoking cessation, and c) comparison between a new pharmacotherapeutic agent and TNP in women.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45. Individuals over the age of 45 will not be included as we are examining the effects of menstrual cycle and ovarian hormones.
* Daily smokers who smoke at least 10 cigarettes per day for at least past 6 months.
* Post menarche and pre menopausal
* Regular menstrual cycle between 25 and 35 days
* At least three months post delivery and breast feeding
* Desire to quit smoking and willingness to participate in a research study.
* Women with a history of depression (but not current MDE) and current PMDD will be included. Excluding women with these diagnoses would have a major impact on feasibility, but because both disorders might impact treatment outcome, individuals will be stratified across randomization groups.

Exclusion Criteria:

* Any unstable major axis I psychiatric disorder in the past month
* Current substance use disorders other than nicotine and caffeine use, in the past 30 days.
* Any medication that may interfere with psychophysiological monitoring
* Unstable medical or serious medical condition in the past 6 months
* Hypersensitivity to varenicline or TNP
* Use of other tobacco products
* Use of other medications with smoking cessation efficacy within 30 days prior to enrollment
* BMI less than 15 since this could alter hormone levels that affect menstrual phase
* Pregnancy
* Breast feeding
* Status post hysterectomy
* Birth control or HRT medication that would effect the menstrual cycle. Currently available oral contraceptives contain either a combination of a synthetic estrogen and synthetic progestin, or a progestin alone. Estrogen and/or progestin inhibit ovulation and alter cervical mucus and the endometrium by suppressing the production of follicle-stimulating hormone and the luteinizing hormone surge (Bucci & Carson, 1997)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2007-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Gray, MD, Principal Investigator — Medical University of South Carolina; Michael E Saladin, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Saladin ME, McClure EA, Baker NL, Carpenter MJ, Ramakrishnan V, Hartwell KJ, Gray KM. Increasing progesterone levels are associated with smoking abstinence among free-cycling women smokers who receive brief pharmacotherapy. Nicotine Tob Res. 2015 Apr;17(4):398-406. doi: 10.1093/ntr/ntu262. PMID 25762749
- [Derived] Gray KM, McClure EA, Baker NL, Hartwell KJ, Carpenter MJ, Saladin ME. An exploratory short-term double-blind randomized trial of varenicline versus nicotine patch for smoking cessation in women. Addiction. 2015 Jun;110(6):1027-34. doi: 10.1111/add.12895. Epub 2015 Mar 29. PMID 25727442

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline: Participant randomized to receive active varenicline and placebo transdermal nicotine patch.
  varenicline: Day -7 thru -5: 0.5mg QD Day -4 thru -1: 0.5mg BID Day 0 onward: 1.0mg BID
  Varenicline is taken for a duration of 4 weeks in this study.
- Transdermal Nicotine Patch: Participant randomized to receive active transdermal nicotine patch and placebo varenicline.
  transdermal nicotine patch: Weeks 0-3: 21mg patch
  Transdermal nicotine patch is used for a duration of 3 weeks in this study.
Period: Overall Study
Arm/Group | Varenicline | Transdermal Nicotine Patch
Started | 67 | 73
Completed | 67 | 73
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Transdermal Nicotine Patch | Total
Number analyzed (Participants) | 67 | 73 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (7.9) | 33.0 (7.4) | 31.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 73 | 140
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 16 | 30
  White | 53 | 57 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: End-of-treatment Abstinence
Description: Carbon monoxide (≤10 parts per million) verified abstinence during the last two weeks of treatment
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Transdermal Nicotine Patch
Number analyzed (Participants) | 67 | 73
Participants | 25 | 13
Statistical Analysis 1: Comparison: Varenicline vs Transdermal Nicotine Patch; Test type: Superiority; p = 0.011, Regression, Logistic; Odds Ratio (OR) = 2.77, 95% CI 2-sided [1.17 to 6.59]

ADVERSE EVENTS:
Arm/Group | Varenicline | Transdermal Nicotine Patch
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/67 | 1/73
Other Adverse Events (participants affected / at risk) | 67/67 | 73/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=67) | Transdermal Nicotine Patch (N=73)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Generalized rash not near patch site
Fever (Infections and infestations) | 0 (0) | 1 (1) — Fever, which accompanied rash
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=67) | Transdermal Nicotine Patch (N=73)
All (Investigations) | 67 (137) | 73 (170)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No